CLINICAL TRIAL: NCT06372405
Title: Instructed Cognitive Reappraisal in Reducing Affective, Behavioral and Psychophysiological Symptoms of Misophonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warsaw, Poland (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSP-501/D125/79/00000
Record Dates: First submitted 2024-03-25; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Misophonia Treatment
Keywords: misophonia; sound over-responsivity; cognitive reappraisal; relaxation training; CBT; psychotherapy; psychophysiology
MeSH Terms: conditions — misophonia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Reappraisal (Experimental): Cognitive reappraisal is a psychotherapeutic strategy utilized to regulate emotions by reinterpreting the meaning of stimuli. Participants will receive instructions on generating and implementing cognitive reappraisal in both misophonic and non-misophonic contexts and will be practicing it within psychotherapeutic sessions. The program consists of four weekly online psychotherapeutic sessions: the first session will be a 90-minute group session, followed by three individual sessions, each lasting 30 minutes.
  Interventions: Behavioral: Cognitive reappraisal
- Schultz Autogenic Training (Active Comparator): Schultz Autogenic Training is a relaxation technique aimed at promoting relaxation and reducing physiological arousal. It consists of six exercises focusing on sensations of heaviness, warmth, heartbeat, breathing, abdominal warmth, and coolness of the forehead.
  Interventions: Behavioral: Schultz Autogenic Training

INTERVENTIONS:
Behavioral: Cognitive reappraisal — Cognitive reappraisal is a psychotherapeutic strategy utilized to regulate emotions by reinterpreting the meaning of stimuli. Participants will receive instructions on generating and implementing cognitive reappraisal (distancing and reframing) in both misophonic and non-misophonic contexts and will be practicing it within psychotherapeutic sessions. The program consists of four weekly online psychotherapeutic sessions: the first session will be a 90-minute group session, followed by three individual sessions, each lasting 30 minutes.
  Arms: Cognitive Reappraisal
Behavioral: Schultz Autogenic Training — Schultz Autogenic Training is a relaxation technique aimed at promoting relaxation and reducing physiological arousal. It consists of six exercises focusing on sensations of heaviness, warmth, heartbeat, breathing, abdominal warmth, and coolness of the forehead. The program consists of four weekly online psychotherapeutic sessions: the first session will be a 90-minute group session, followed by three individual sessions, each lasting 30 minutes.
  Arms: Schultz Autogenic Training

SUMMARY:
Misophonia is a disorder causing intense reactions to specific sounds, disrupting daily life. Current treatments lack evidence-based support. The goal of this study is to explore the effectiveness of cognitive reappraisal (CR) in reducing misophonic responses. The study involves 100 participants assigned to either a 4-week CR program or Autogenic Training. Emotional regulation, symptoms of anxiety and depression, quality of life, and more will be assessed using various questionnaire-based measures; perseverations with a task-based test (Wisconsin Card Sorting Test); the presence of psychiatric and personality disorders using face-to-face interviews (The Mini-International Neuropsychiatric Interview (M.I.N.I.) and "Structured Clinical Interview for DSM-5® Personality Disorders" (SCID-5-PD)

DETAILED DESCRIPTION:
Misophonia is a condition characterized by a reduced tolerance for certain repetitive stimuli, particularly sounds, leading to significant disruptions in daily functioning. Despite ongoing efforts to understand its mechanisms and develop effective treatments, there is currently no established intervention for misophonia. While preliminary research suggests cognitive reappraisal (CR) might help with misophonia symptoms, no studies have directly investigated its effectiveness in individuals with misophonia.

Our main goal is to assess how effective brief instructed CR and a 4-week CR training program are in regulating emotional responses among individuals with misophonia. ]The following outcomes are anticipated:

1. After completing a dedicated 4-week CR program targeting misophonia, participants are expected to exhibit improved emotional regulation in response to misophonic triggers. This improvement should lead to reduced misophonia symptoms, particularly noticeable in experimental tasks involving misophonic triggers and in questionnaire-based assessments, especially in the Externalizing and Impact (S-Five) scales. In the active control group (AT), the investigators predict no change in emotional response (Manikin scales) in the experimental task responses to misophonic and non-misophonic triggers. Additionally, the investigators expect no decrease in misophonia symptoms in the Externalizing Scale based on questionnaire assessments. However, in the control group (AT), a slight, but not significant, reduction in overall misophonia, anxiety, and depression symptoms is anticipated, reflected in questionnaire assessments.
2. Participants may regulate emotional responses less effectively using CR in response to misophonia-specific aversive stimuli compared to non-misophonia-related aversive stimuli, both before and after the misophonia-focused 4-week CR training.
3. The misophonia-focused 4-week CR training will significantly enhance the effectiveness of short cognitive reappraisal training.

Additionally, the investigators aim to explore factors that might affect intervention outcomes, such as comorbid disorders, perseveration, relationship with the therapist during CR training, attitudes towards the treatment, and more.

EXPERIMENTAL ASSESSMENT The experimental assessment in the psychophysiology lab aims to evaluate the ability to use instructed cognitive reappraisal before and after four weeks of training. Before the experiment, there will be a 10-minute instruction session to teach the participants (in CR group) this technique. During the experiment, participants will be presented with a series of misophonic (3), non-misophonic aversive stimuli (3), and neutral stimuli (3), each lasting 30 seconds; presented in quasi-randomized balanced orders. The aversive (misophonia and non-misophonic) audio-video stimuli will be presented under two conditions: 'look', where participants will be instructed to only look and not use any strategies to regulate their emotions, and 'decrease', where they will have to use a cognitive reappraisal (CR) technique to decrease their unpleasant emotions/arousal (or 'trying to think in a way to decrease the unpleasant emotions' in the control group). The neutral conditions will also be presented twice each, but always with the instruction 'look'. After each stimulus presentation, participants will be asked to rate their emotions using the Manikin scales for valence and arousal. At the end of the trials, they will be asked to report the amount of effort (on a 10-point scale) they had to exert for each of the aversive stimuli. Physiological data (heart rate (HR), Skin Conductance Response (SCR), and facial corrugator by electromyography (EMG) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification of experiencing stress due to eating sounds, confirmed during a subsequent online face-to-face diagnostic meeting,
* Confirmation of misophonia symptoms through a face-to-face/online interview using the Duke Misophonia Interview (DMI; Polish adaptation),
* being fluent in the Polish language,
* age range: 18-55,
* not having been in therapy within the last 3 months.

Exclusion Criteria:

* Individuals identified with misophonia (indicated by DMI) who do not experience triggers related to eating sounds,
* At the time of recruitment: individuals meeting criteria for current mania, anorexia, psychotic episode/disorder, significant or sudden crisis, or reporting current suicidal ideations,
* Individuals with heart diseases or pacemakers, or those taking cardiac medications,
* Individuals reporting a diagnosis of hearing loss or significant hearing difficulties.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in misophonia symptoms measured by S-Five - Externalizing subscale | 1st assessment - 3-10 days before the 1st therapy session. 2nd assessment: 3-10 days after the last (the 4th) therapy session. (There are 4 weekly sessions throughout one month).
  S-Five is a validated questionnaire used in Poland to assess misophonia symptoms. Higher values indicate more severe misophonia symptoms, with a range of 0-50 for each subscale.
Change in misophonia symptoms measured by S-Five - Internalizing subscale | 1st assessment - 3-10 days before the 1st therapy session. 2nd assessment: 3-10 days after the last (the 4th) therapy session. (There are 4 weekly sessions throughout one month).
  S-Five is a validated questionnaire used in Poland to assess misophonia symptoms. Higher values indicate more severe misophonia symptoms, with a range of 0-50 for each subscale.
Change in misophonia symptoms measured by S-Five - Threat subscale | 1st assessment - 3-10 days before the 1st therapy session. 2nd assessment: 3-10 days after the last (the 4th) therapy session. (There are 4 weekly sessions throughout one month).
  S-Five is a validated questionnaire used in Poland to assess misophonia symptoms. Higher values indicate more severe misophonia symptoms, with a range of 0-50 for each subscale.
Change in misophonia symptoms measured by S-Five - Impact subscale | 1st assessment - 3-10 days before the 1st therapy session. 2nd assessment: 3-10 days after the last (the 4th) therapy session. (There are 4 weekly sessions throughout one month).
  S-Five is a validated questionnaire used in Poland to assess misophonia symptoms. Higher values indicate more severe misophonia symptoms, with a range of 0-50 for each subscale.
CHange in misophonia symptoms measured by S-Five - Outburst subscale | 1st assessment - 3-10 days before the 1st therapy session. 2nd assessment: 3-10 days after the last (the 4th) therapy session. (There are 4 weekly sessions throughout one month).
  S-Five is a validated questionnaire used in Poland to assess misophonia symptoms. Higher values indicate more severe misophonia symptoms, with a range of 0-50 for each subscale.
Change of aversiveness rating (valence/pleasure) on the Manikin Scales. | 1st assessment - 3-8 days before the 1st therapy session. 2nd assessment: 3-8 days after the last (the 4th) therapy session. (There are 4 weekly sessions throughout one month).
  Manikin Scales are commonly used scales to assess emotional valence. Range: 1-5. Higher values indicate higher aversiveness/lower pleasure.
  A change in ratings during the 'decrease' condition, compared to the 'look' condition is expected. This change is expected to be more pronounced in the post-treatment assessment than at the baseline assessment (before therapy), particularly regarding misophonic triggers. No changes are anticipated in the control group.
Change of arousal rating on the Manikin Scales. | 1st assessment - 3-8 days before the 1st therapy session. 2nd assessment: 3-8 days after the last (the 4th) therapy session. (There are 4 weekly sessions throughout one month).
  Manikin Scales are commonly used scales to assess emotional valence. Range: 1-5. Higher values indicate lower arousal.
  A change in ratings during the 'decrease' condition, compared to the 'look' condition is expected. This change is expected to be more pronounced in the post-treatment assessment than at the baseline assessment (before therapy), particularly regarding misophonic triggers. No changes are anticipated in the control group.
Change in Galvanic Skin Response | 1st assessment - 3-8 days before the 1st therapy session. 2nd assessment: 3-8 days after the last (the 4th) therapy session. (There are 4 weekly sessions throughout one month).
  Higher values here indicate arousal linked to misophonic reactions/higher misophnic reaction.
Change in average HR during the trigger presentation | Baseline vs. post-treatment assessment (which will be performed 5 to 12 weeks since the last session).
  Higher values here indicate arousal linked to misophonic reactions/higher misophnic reaction.
Diagnosis of personality disorders as a predictor of worse treatment outcome. | 3 to 10 days before the 1st session
  Personality disorders will be assessed using the SCID-5-PD (Polish adaptation). It is anticipated that meeting the criteria for a PD (especially higher symptoms OCPD) will be related to poorer treatment outcomes.
Working Alliance Inventory will be related to better treatment outcomes. | 3-8 days after the last (the 4th) therapy session (There are 4 weekly sessions throughout one month)
  Higher scores indicate a better quality of relationship with therapist. Range: 12-84.

SECONDARY OUTCOMES:
Meeting criteria for psychiatric disorders - | 3 to 10 days before the 1st session
  Psychiatric disorders will be assessed using a structured interview - the Mini International Neuropsychiatric Interview (Polish adaptation). It is anticipated that meeting the criteria for at least one psychiatric disorder will correlate with higher misophonia symptoms and worse treatment outcomes.
Hearing test - standard and high frequency pure-tone audiometry | 3 to 10 days after the 4st session
  It is predicted that the results of pure-tone audiometry will not be related to either the severity of misophonia symptoms or the treatment outcome. The standard audiometry range is 250Hz to 8kHz, while high-frequency audiometry covers the range from 10kHz to 20kHz.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Psychology, University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided